CLINICAL TRIAL: NCT05762848
Title: Clinical Application and Functionality for an Application for Measurement of Head Circumference in Neonates and Children
Brief Title: Clinical Application and Functionality for an Application for Measurement of Head Circumference.
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Mr Stefan Yordanov, Research Neurosurgical Registrar, University of Cambridge
Other Study IDs: Ver2
Record Dates: First submitted 2022-05-16; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Hydrocephalus in Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Researcher: Patients will have their Head circumference measured with a tape and with the mobile phone app.
  Interventions: Device: Mobile Phone Head Circumference App
- Parent: Patients will have their Head circumference measured with a tape and with the mobile phone app.
  Interventions: Device: Mobile Phone Head Circumference App

INTERVENTIONS:
Device: Mobile Phone Head Circumference App — Measurement of Head circumference of Babies/Infants with a mobile phone application.

SUMMARY:
Title of clinical study:Clinical application, validation, and functionality evaluation of the Mobile Head Circumference Application in neonates and children

Sponsor: University Hospitals NHS Foundation Trust

Purpose of study:Evaluate and validate the utility of the mobile Head Circumference application for use in the clinical and outpatient setting for evaluation of head circumference of neonates and infants

Primary objectives:Evaluate usefulness of and feasibility of the application in the clinical setting comparing it to normal practice.

Secondary objectives:Evaluate parent/guardian reliability and satisfaction of the use of the mobile head circumference app.

Study Design:Prospective

Sample Size:Treating clinicians employed by Cambridge University Hospitals NHS Foundation Trust will identify patients eligible for this study (infants <18 months of age) and notify research team members with the patient's/guardian's consent. Once identified, research team members will approach patients' parents/guardians to seek informed consent before their clinic appointment or at the bedside on the ward. An information sheet will be used. If they choose to participate, we will measure the HC during the clinic appointment or on the ward. (Please refer to Flowchart 1). Sample size estimation was calculated with 90% statistical power to detect a change of means by 1 and a standard deviation of 1. This, along with 10% iteration, equals 33 participants.

Summary of eligibility criteria:Neonatal patients and infants with need of continuous measurement of Head Circumference up to the age of 18months.

Investigational techniques:Mobile application for Automatic measurement of head circumference.

DETAILED DESCRIPTION:
An accurate head circumference (HC) measurement is a quick and cost-effective assessment which is essential when clinically evaluating a neonate or infant. HC outside the normal range may indicate a disorder of brain development, hydrocephalus, or an intracranial mass lesion. The growth pattern of HC, determined from serial measurements, also provides useful clinical information. For example, changes in HC are used to help determine whether hydrocephalus needs treatment. HC growth is also predictive of neurodevelopmental outcomes. [Lippé et al. 2018]

HC is measured by measuring the widest circumference of the head with a tape measure. Typically, this is performed by health care workers, but parents can be taught to take measurements reliably. With the increasing use of telephone and virtual clinics as a substitute to face-to-face appointments, parental measurement of HC is increasingly used to help guide clinical management in a wide variety of clinical specialties including Neurosurgery, Neonatology, Paediatrics, and General Practice.

Tape measure HC measurements are prone to error, particularly when performed by parents, due to individual differences in head shape, hair style and texture, subject cooperation, and examiner differences in tape measure placement and tautness.6 There is therefore the need for a more reliable method.

Rationale for the study:

We have developed a HC mobile application (HCMA) that can measure the head circumference of an infant and plot it against standardised growth charts.

The rationale of this study is to validate the HCMA in a clinical setting and to review its usability by parents in the community.

Research objective and purpose

The main objective of the study is to validate the accuracy of the HC app and to prove its utility and feasibility in clinical practice.

Secondary objectives will be to evaluate parent/guardian reliability and satisfaction of using the HC app.

Primary Objective:

Hypothesis 1: There is no statistically significant difference between HC measured with a tape measure and HC measured with HCMA;

Secondary Objectives:

Hypothesis 2: Intra-rater Reliability(precision/repeatability) - The variability of series of three measurements of HC using HCMA (performed by a healthcare professional) is within 0.5 cm -(the standard error margin for measurement measurements) Hypothesis 3: Inter-rater Reproducibility - HC measurements made using the HCMA will not be significantly different when measured by parents or healthcare professionals we will then compare measurements of HC using HCMA performed by healthcare professional with the measurements performed by the parents/guardians using the HCMA. These should be within the standard error of margin for the measurement with tape measure.

Hypothesis 4: Parents are satisfied using the HCMA and find it easy to use'

ELIGIBILITY:
Inclusion Criteria:

* Infants up to 18 months old seen in a paediatric clinic with a requirement for continuous head circumference measurements.

Exclusion Criteria:

* Infants above the age of 18 months, Patients in emergency setting, Withdrawal of consent of parents/guardians

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants up to 18 months with neurological disorders(attending Neurosurgery Clinics)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Criterion Validity(Vs Gold Standard) | Day 0
  Proof of concept of that the HCMA is an accurate and precise tool for measuring HC compared to standard practice (tape measure);

SECONDARY OUTCOMES:
Repeatability and reliability | Day 0
  Within-rater variability using three consecutive measurements with HCMA by a health care professional;
Reliability of parents/guardians in measurement of head circumference with a tape measure (supervised by a health care professional); | Day 0
Reliability of parents/guardians in measurement of head circumference using the HCMA | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Jalloh, FRCS(Nsgy), Principal Investigator — University of Cambridge; Stefan Yordanov, MRCSed, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Cole TJ, Freeman JV, Preece MA. British 1990 growth reference centiles for weight, height, body mass index and head circumference fitted by maximum penalized likelihood. Stat Med. 1998 Feb 28;17(4):407-29. PMID 9496720
- [Result] Dupont C, Castellanos-Ryan N, Seguin JR, Muckle G, Simard MN, Shapiro GD, Herba CM, Fraser WD, Lippe S. The Predictive Value of Head Circumference Growth during the First Year of Life on Early Child Traits. Sci Rep. 2018 Jun 29;8(1):9828. doi: 10.1038/s41598-018-28165-8. PMID 29959368
- [Result] Engle WA; American Academy of Pediatrics Committee on Fetus and Newborn. Age terminology during the perinatal period. Pediatrics. 2004 Nov;114(5):1362-4. doi: 10.1542/peds.2004-1915. PMID 15520122
- [Result] Sullivan JC, Tavassoli T, Armstrong K, Baron-Cohen S, Humphrey A. Reliability of self, parental, and researcher measurements of head circumference. Mol Autism. 2014 Jan 10;5(1):2. doi: 10.1186/2040-2392-5-2. PMID 24410855